CLINICAL TRIAL: NCT02975895
Title: Outcome With Hydrophobic and Hydrophilic Intraocular Lens in Patients With and Without Uveitis
Brief Title: Outcome of Different IOLs in Patients With and Without Uveitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 031-16
Record Dates: First submitted 2016-11-15; First posted 2016-11-29 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Uveitis; Cataract; Inflammation; Posterior Capsule Opacification
MeSH Terms: conditions — Uveitis; Cataract; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrophobic IOL: Vivinex (HOYA) (Other): Intraocular lens with hydrophobic properties: Vivinex (HOYA).
  Interventions: Device: Hydrophobic IOL: Vivinex (HOYA)
- Hydrophilic IOL: INCISE (Bausch+Lomb) (Other): Intraocular lens with hydrophilic properties: INCISE (Bausch+Lomb).
  Interventions: Device: Hydrophilic IOL: INCISE (Bausch+Lomb)

INTERVENTIONS:
Device: Hydrophobic IOL: Vivinex (HOYA) — Patients requiring cataract surgery will be randomized to one of the two types of IOLs.
  Arms: Hydrophobic IOL: Vivinex (HOYA)
Device: Hydrophilic IOL: INCISE (Bausch+Lomb) — Patients requiring cataract surgery will be randomized to one of the two types of IOLs.
  Arms: Hydrophilic IOL: INCISE (Bausch+Lomb)

SUMMARY:
Cataract, is a clouding of the lens in the eye gradually leading to reduction of the visual acuity. In most cases it can be managed with surgery, removing the own lens and replacing it with an artificial lens, intraocular lens (IOL). These lenses are made in different materials with different properties.

Uveitis refers to an inflammation in the iris, ciliary body and choroid. Patients with this disease have an increased risk of developing cataract due to the inflammation itself and treatment with steroids. They also have an increased risk of complications during surgery and postoperatively. In this group the selection of IOL might be of greater importance.

The aim of this prospective randomized controlled study is to compare the outcome of hydrophobic and hydrophilic intraocular lenses in patients with and without uveitis

ELIGIBILITY:
Inclusion Criteria:

* Cataract requiring surgery
* Ability to understand and sign consent form

Exclusion Criteria:

* Extensive corneal scarring
* Other eye surgery less than 3 months before inclusion
* Unregulated glaucoma
* Active uveitis (increased inflammation and treatment less than 3 months before inclusion)
* Intraoperative complications (capsular tear or vitreous loss)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory response | Preoperatively and at seven occasions within two years postoperatively

SECONDARY OUTCOMES:
Evaluation of posterior capsule opacification after six months | Six months (plus or minus 30 days) postoperatively
Evaluation of posterior capsule opacification after one year | One year (plus or minus 30 days) postoperatively
Evaluation of posterior capsule opacification after two years | Two years (plus or minus 2 months) postoperatively
Change in best corrected visual acuity assessed in decimal using Snellen charts | Preoperatively and at six occasions within two years postoperatively
Complications | Preoperatively and at seven occasions within two years postoperatively
  Postoperative glaucoma or cystoid macular edema

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Zetterberg, MD, PhD, Principal Investigator — Västra Götalands regionen, Sahlgrenska University Hospital, Department of Ophthalmology
Locations (1):
- Vastra Gotaland Region, Sahlgrenska University Hospital, Department of Ophthalmology, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: Undecided